CLINICAL TRIAL: NCT00502710
Title: A Randomized, Double-blind Dose-ranging Study of the Effect of DPP-IV on HbA1c, Other Efficacy Parameters, Pharmacokinetics and Safety in Patients With Type 2 Diabetes (BC20779)
Brief Title: A Study of Dipeptidyl-peptidase IV (DPP-IV) RO4876904 in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20779
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- RO4876904 1 (Experimental): Escalating doses, at a starting dose of 12.5mg po daily. Patients receiving metformin before the study will continue on the same dose of metformin.
  Interventions: Drug: RO4876904
- RO4876904 2 (Experimental): Escalating doses, at a starting dose of 12.5mg po daily. Patients receiving metformin before the study will continue on the same dose of metformin.
  Interventions: Drug: RO4876904
- RO4876904 3 (Experimental): Escalating doses, at a starting dose of 12.5mg po daily. Patients receiving metformin before the study will continue on the same dose of metformin.
  Interventions: Drug: RO4876904
- RO4876904 4 (Experimental): Escalating doses, at a starting dose of 12.5mg po daily. Patients receiving metformin before the study will continue on the same dose of metformin.
  Interventions: Drug: RO4876904
- Placebo (Placebo Comparator): Placebo po daily. Patients receiving metformin before the study will continue on the same dose of metformin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo po daily.
  Arms: Placebo
Drug: RO4876904 — Escalating doses, at a starting dose of 12.5mg po daily.
  Arms: RO4876904 1; RO4876904 2; RO4876904 3; RO4876904 4

SUMMARY:
This 5 arm study will assess the efficacy, pharmacokinetics, safety and tolerability of a DPP-IV inhibitor compared to placebo in patients with type 2 diabetes. Patients will be randomized to receive DPP-IV(3) at one of 4 doses (of 12.5mg and above), or placebo p.o. Patients receiving metformin before the study will continue on the same dose of metformin. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes diagnosed >= 1 month before screening;
* drug-naive, or pretreated with maximum tolerated dose (MTD) of metformin;
* BMI 25-45kg/m2.

Exclusion Criteria:

* type 1 diabetes;
* any anti-hyperglycemic medication other than metformin, or weight-lowering drug, during last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Absolute change in hemoglobin A1c (HbA1c) | Week 12

SECONDARY OUTCOMES:
Absolute change in fasting plasma glucose (FPG), HbA1c response rate, absolute/relative change in insulin sensitivity, beta cell function, lipid profile. | Week 12
Adverse events (AEs), vital signs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (12):
  - Hot Springs, Arkansas
  - Concord, California
  - Los Angeles, California
  - Chicago, Illinois
  - Avon, Indiana
  - Indianapolis, Indiana
  - Oxon Hill, Maryland
  - Troy, Michigan
  - Omaha, Nebraska
  - Binghamton, New York
  - Charlotte, North Carolina
  - Beaver, Pennsylvania
- Australia (3):
  - Adelaide
  - Canberra
  - St Leonards
- São Paulo, Brazil
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Mexico (6):
  - Aguascalientes
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - Pachuca
  - Tampico
- Russia (4):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Spain (5):
  - Alzira
  - Bacarot Alicant
  - Badalona
  - Barcelona
  - Ferrol
- United Kingdom (5):
  - Bath
  - Frome
  - Glasgow
  - Liverpool
  - Motherwell